CLINICAL TRIAL: NCT06685718
Title: Phase 1a/1b, Open-Label Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of a CDAC Degrading EGFR, BG-60366, in Patients With EGFR-Mutant Non-Small Cell Lung Cancer
Brief Title: A Study Investigating BG-60366 in Adults With Epidermal Growth Factor Receptor (EGFR)-Mutant Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-60366-101; 2024-517322-26-00 (EU CTIS Number); CTR20250272 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Lung Cancer; NSCLC; NSCLC (Non-small Cell Lung Carcinoma); EGFR Activating Mutation; EGFR Mutation-Related Tumors
Keywords: lung cancer; non-small cell lung cancer; NSCLC; EGFR activating mutation; EGFR resistant mutation; advanced or metastatic non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation and Safety Expansion (Experimental): Sequential cohorts of increasing dose levels of BG-60366 will be evaluated as monotherapy.
  Interventions: Drug: BG-60366
- Phase 1b: Dose Expansion (Experimental): Recommended Dose(s) for Expansion (RDFE[s]) of BG-60366 as monotherapy determined from Phase 1a will be evaluated.
  Interventions: Drug: BG-60366

INTERVENTIONS:
Drug: BG-60366 — Administered orally

SUMMARY:
This is an open-label, multicenter, Phase 1a/1b clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of BG-60366, a highly potent, selective EGFR-mutation targeted Chimeric Degradation Activation Compound (CDAC). BG-60366 is designed to degrade mutant EGFR, which is a common cause for Non-Small Cell Lung Cancer (NSCLC). This study will evaluate how well BG-60366 works in participants with advanced or metastatic EGFR-mutant NSCLC.

The study will be conducted in 2 parts: 1) Phase 1a Dose Escalation and Safety Expansion, and 2) Phase 1b Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC, carrying an EGFR activating mutation prior to receiving standard EGFR-tyrosine kinase inhibitor (EGFR-TKI)
* Phase 1a general inclusion criteria:

  * Disease progression on prior third-generation EGFR-TKI for advanced or metastatic disease, and either progressed or ineligible for currently available standard-of-care treatment (eg, platinum-based chemotherapy) after EGFR-TKI treatment
* Phase 1a safety expansion

  * Documentation of EGFR resistance mutations (ie, C797s)
* At least ≥ 1 evaluable lesion (for Phase 1a Dose Escalation) or at least ≥ 1 measurable lesion (for Phase 1a Safety Expansion or Phase 1b Dose Expansion) per RECIST v1.1
* EGFR resistance mutations may be detected locally either from tumor tissue or circulating tumor DNA (ctDNA) in blood, and samples used for detection of resistance mutations must be collected after progression on the most recent systemic antitumor treatment
* Adequate organ function
* Stable Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1

Exclusion Criteria:

* Any previous histologic or cytologic evidence of small cell or combined small cell/non-small cell disease in the archival tumor tissue or tumor biopsy before enrollment
* Symptomatic spinal cord compression
* Brain metastases which are symptomatic and/or requiring emergency treatment (eg, starting steroid, or stereotactic radiation/whole-brain radiation within 2 weeks before first dose of study drug)
* Prior treatment with fourth-generation EGFR-TKI, other CDAC/proteolysis-targeting chimeras (PROTAC) compounds targeting EGFR mutations, or other drugs with the mechanism of action specifically targeting EGFR resistance mutations (eg, C797X) (except for the first- to third-generation EGFR-TKIs)
* Any history of interstitial lung disease (ILD) or ≥ Grade 2 noninfectious pneumonitis ≤ 2 years before the first dose of study drug, or has current ILD/noninfectious pneumonitis, or where suspected active ILD/noninfectious pneumonitis cannot be ruled out by imaging during screening
* Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose of the study drug to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first (approximately 18 months)
  Number of participants with AEs and SAEs, including findings from laboratory assessments, electrocardiograms (ECGs), and physical examinations, and that meet protocol-defined dose-limiting toxicity (DLT) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) | Approximately 1 month
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended dose(s) for expansion (RDFE) of BG-60366 | Approximately 18 months
  RDFE of BG-60366 will be determined based upon the MTD or MAD.
Phase 1b: Number of Participants with Adverse Events and Serious Adverse Events | From first dose of the study drug to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first (approximately 24 months)
  Number of participants with AEs and SAEs, including findings from physical examinations, ECGs, and laboratory assessments as needed.
Phase 1b: Overall Response Rate (ORR) | Approximately 24 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1a: Overall Response Rate (ORR) | Approximately 24 months
  ORR is defined as the percentage of participants who had confirmed CR or PR assessed by the investigator using RECIST v1.1.
Phase 1a and 1b: Duration of Response (DOR) | Approximately 24 months
  DOR is defined as the time from the first determination of objective response that is confirmed by the subsequent assessment until the first documentation of disease progression or death, whichever comes first.
Phase 1a and 1b: Time to Response (TTR) | Approximately 24 months
  TTR is defined as the time from the date of the first dose of study drugs to the date of teh first determination of objective response that is confirmed by the subsequent assessment.
Phase 1b: Progression-Free Survival (PFS) | Approximately 24 months
  PFS is defined as the time from the date of the first dose of study drug to the date of the first documentation of disease progression assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Disease Control Rate (DCR) | Approximately 24 months
  DCR is defined as the percentage of participants with the best overall response of confirmed CR, PR, or stable disease assessed.
Phase 1a and 1b: Maximum observed plasma concentration (Cmax) of BG-60366 | Twice in the first 3 months
Phase 1a and 1b: Time to reach maximum observed plasma concentration (Tmax) of BG-60366 | Twice in the first 3 months
Phase 1a and 1b: Apparent terminal elimination half-life (t1/2) of BG-60366 | Twice in the first 3 months
Phase 1a and 1b: Area under the concentration-time curve (AUC) for BG-60366 | Twice in the first 3 months
Phase 1a and 1b: Minimum observed plasma concentration (Cmin) of BG-60366 | Twice in the first 3 months
Phase 1a and 1b: Apparent total clearance (CL/F) of BG-60366 | Twice in the first 3 months
Phase 1a and 1b: Apparent volume of distribution (Vz/F) of BG-60366 | Twice in the first 3 months
Phase 1a and 1b: Accumulation Ratio (AR) of BG-60366 | Once in the first three months
Phase 1a and 1b: Plasma concentrations of BG-60366 | Approximately up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (28):
- United States (6):
  - University of Colorado, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Ohio State University, Columbus, Ohio
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital Huifu Branch, Guangzhou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical Universitywuxiang Branch, Nanning, Guangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicineqiantang Branch, Hangzhou, Zhejiang
- Italy (2):
  - Fondazione Irccs San Gerardo Dei Tintori Sc Oncologia, Monza
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Harbour Cancer and Wellness, Auckland, New Zealand
- South Korea (3):
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (3):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Hospital Universitario de Octubre, Madrid
  - H Puerta de Hierro Majadahonda, Majadahonda

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/